CLINICAL TRIAL: NCT04321304
Title: Impact of Transcranial Direct Current Stimulation Intensity on Leg Muscle Fatigability in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Craig D. Workman, PhD, Postdoctoral Scholar, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201902799
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: Brain Stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham (Sham Comparator): Participants will have the anode (active electrode) placed over the brain area the controls their dominant leg and the cathode (return electrode) above the ipsilateral eyebrow. Stimulation is turned on (2 mA) for the 30 seconds at the beginning and the end of the trial, but stays at 0 mA in the intervening time.
  Interventions: Device: Sham transcranial direct current stimulation
- 2 mA (Experimental): Participants will have the anode (active electrode) placed over the brain area the controls their dominant leg and the cathode (return electrode) above the ipsilateral eyebrow. Stimulation is ramped up to 2 mA over the first 30 seconds and stays at 2 mA for the remainder of the stimulation time.
  Interventions: Device: Transcranial direct current stimulation at 2 mA
- 4 mA (Experimental): Participants will have the anode (active electrode) placed over the brain area the controls their dominant leg and the cathode (return electrode) above the ipsilateral eyebrow. Stimulation is ramped up to 4 mA over the first 30 seconds and stays at 4 mA for the remainder of the stimulation time.
  Interventions: Device: Transcranial direct current stimulation at 4 mA

INTERVENTIONS:
Device: Sham transcranial direct current stimulation — Uses weak electrical current (2 mA intensity) at the beginning and the end of a given stimulation period to control for potential placebo-like effects or participant expectation bias.
  Other Names: tDCS
  Arms: Sham
Device: Transcranial direct current stimulation at 2 mA — Uses weak electrical current (2 mA intensity) to either increase or decrease brain excitability and improve functional or cognitive outcomes.
  Arms: 2 mA
Device: Transcranial direct current stimulation at 4 mA — Uses weak electrical current (4 mA intensity) to either increase or decrease brain excitability and improve functional or cognitive outcomes.
  Arms: 4 mA

SUMMARY:
Transcranial direct current stimulation (tDCS) is a painless,non-invasive means of increasing brain excitability. It has been used for several years and in many populations to improve physical and psychological outcomes. Although many tDCS devices are capable of a range of stimulation intensities (e.g., 0 mA - 5 mA), the intensities currently employed in most tDCS research are ≤ 2 mA, which are sufficient to elicit measurable improvements; but, these improvements might be expanded at higher intensities. In the beginning, when the safety of tDCS was still being established for human subjects, careful and moderate approaches to stimulation protocols were warranted. However, recent work using stimulation at higher intensities, i.e. up to 4 mA, has been performed in many populations and was found to have no additional negative side-effects. Now that the safety of tDCS at higher intensities is better established, work exploring the differences in performance between moderate (i.e. 2 mA) and higher (i.e. 4 mA) intensities is necessary to determine if increasing intensity increases the effectiveness of the desired outcome.

Prospective participants will include 40 healthy young adults (all right-side dominant) that will be recruited to complete four randomly ordered stimulation sessions (Baseline, 2 mA, 4 mA, and sham), separated by at least 5 days. Each session will involve one visit to the Integrative Neurophysiology Laboratory (INPL) and will last for approximately one hour. We expect data collection to last 6 months. The first session includes leg strength measurements and fatigue tasks of both legs, as well as a baseline 6 min walk test (6MWT) to determine fatigued walking characteristics. The following three sessions will include performing a random tDCS condition (2 mA, 4 mA, or sham) over the brain area that controls the participant's dominant leg for 15 minutes prior to and then throughout the duration of the fatigue task of the dominant leg (16-20 min total stimulation time). The fatigue task for the nondominant leg will be performed after a 10 minute energy recovery period. After the fatigue task has been completed for both legs, the participants will perform the 6MWT.

ELIGIBILITY:
Inclusion Criteria:

1. Young adult (18-30 yrs)
2. right-side dominant
3. able to independently walk for 6 min
4. at least 30 min of moderate-intensity, physical activity on at least 3 days of the week for at least the last 3 months
5. without chronic neurological, psychiatric, or medical conditions
6. not taking any psychoactive medications

Exclusion Criteria:

1. pregnant
2. known holes or fissures in the skull
3. metallic objects or implanted devices in the skull (e.g., metal plate)
4. current student of study personnel
5. under the direct supervision of study personnel

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Distance walked in the 6 Minute Walk Test | Through study completion, up to 6 months
  Walk back and forth between two markers spaced 30 meters apart for six minutes
Fatigue index from the isokinetic fatigue test | Through study completion, up to 6 months
  Perform 40 consecutive flexion and extension repetitions of the knee on the dominant leg. After a 10 minute rest, do the same task on the the non-dominant leg.

CONTACTS AND LOCATIONS:
Overall Officials: Craig D Workman, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States